CLINICAL TRIAL: NCT01107145
Title: A Multi-center, Open-label, Randomized Trial of Chloroquine, Artemether-Lumefantrine, and Mefloquine-Artesunate for the Treatment of Uncomplicated P. Vivax Malaria in Pregnant Women in Brazil
Brief Title: Efficacy of Artemisinin Combination Therapies for the Treatment of Uncomplicated P. Vivax in Pregnancy in Brazil (PAACT-PV)
Acronym: PAACT-PV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Extremely slow enrollment
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAACT-PV
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Plasmodium Vivax Malaria
Keywords: Plasmodium; Vivax; Malaria; Pregnancy; Brazil; Treatment
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — Artemether, Lumefantrine Drug Combination; lactitol; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mefloquine- Artesunate (Experimental): Mefloquine- Artesunate (Farmaguinhos, Brazil): tablets of 100 mg artesunate and 220 mg mefloquine (fixed dose combination), given once daily for 3 days.
  Interventions: Drug: Mefloquine- Artesunate
- Artemether-Lumefantrine (Experimental): Artemether-Lumefantrine, Lumet, Cipla 4 tablets containing 20 mg of artemether plus 120 mg of lumefantrine per tablet twice daily for three days as 2 doses 8 hours apart on the 1st day and then 2 doses 12 hours apart on the 2nd and 3rd days, administered with a fatty meal
  Interventions: Drug: Artemether-Lumefantrine
- Chloroquine (Active Comparator): Chloroquine (Farmaguinhos, Brazil): Tablets containing 250 mg Chloroquine salt given as 4 tablets at once on the first day (or 10 mg/kg) followed by 3 tablets once daily for the next 2 days (or 7,5 mg/kg)
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Mefloquine- Artesunate — Tablets of 100 mg artesunate and 220 mg mefloquine (fixed dose combination), given once daily for 3 days.
  Other Names: Artesunato-Mefloquina (Farmaguinhos, Brazil)
  Arms: Mefloquine- Artesunate
Drug: Artemether-Lumefantrine — 4 tablets containing 20 mg of artemether plus 120 mg of lumefantrine per tablet twice daily for three days as 2 doses 8 hours apart on the 1st day and then 2 doses 12 hours apart on the 2nd and 3rd days, administered with a fatty meal
  Other Names: Coartem, Novartis; Lumet, Cipla
  Arms: Artemether-Lumefantrine
Drug: Chloroquine — Tablets containing 250 mg Chloroquine salt given as 4 tablets at once on the first day (or 10 mg/kg) followed by 3 tablets once daily for the next 2 days (or 7,5 mg/kg)
  Other Names: Chloroquine (Farmaguinhos, Brazil)
  Arms: Chloroquine

SUMMARY:
The current treatment recommendations for P. vivax in pregnant and non-pregnant individuals are to use chloroquine; in non-pregnant patients this is followed by primaquine to prevent relapse. As primaquine can not be used in pregnant women, these women remain at risk of relapse. As there is increasing concern about chloroquine resistant P. vivax in this region, there is a need to identify alternative treatment options. The artemisinin combination therapies are recommended for use against P. falciparum infections in pregnant women after the 1st trimester; additional data are needed to support the use of these drugs against P. vivax.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age >16 weeks (determined by LMP and fundal height)- if there is discordance between the two, the more conservative estimate (i.e. lower) will be used, to prevent accidental exposure of a 1st trimester fetus
* Normal fetal heart beat detected by Doppler
* Presence of asexual P. vivax parasitemia ≤ 50,000 parasites/microliter (thick smear)
* Willing to sign or thumb print informed consent
* Willing to return for scheduled follow up visits for treatment and observation until delivery
* Willing to deliver in health facility

Exclusion Criteria:

* Pregnancy < 16 weeks
* Microscopically confirmed P. falciparum or mixed infection/ parasitemia (P. vivax and another species of Plasmodium, i.e. P. vivax, P. ovale, or P. malariae)
* History of allergy or hypersensitivity to interventional drugs
* Exposure to antimalarial drugs and other drugs with antimalarial activity within the past 2 months, as determined by history from the woman (quinine, mefloquine, or artemisinin derivatives, including AL and MA)
* Patients taking drugs with possible interaction with study drugs (ie. warfarin, digoxin)
* History or family history of epilepsy or psychiatric disorder
* Presence of signs and symptoms of severe malaria, severe illness, or danger signs
* Hemoglobin < 7 g/dl
* Inability to tolerate oral medication (repeated vomiting, impairment of consciousness).
* History of chronic disease including diabetes, renal failure, hepatic failure, heart disease requiring anti-arrhythmic drugs or warfarin, HIV/ AIDS, known hemoglobinopathy
* Participant's inability to return for follow up visits
* Age <15 years

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
63-day PCR-adjusted parasitological cure of P. vivax | 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Meghna Desai, MPH PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- Brazil (3):
  - Hospital Geral Maternidade de Cruzeiro do Sul, Cruzeiro do Sul, Acre
  - Hospital Municipal Teonila Alves, Anajás, Pará
  - Centro de Pesquisa em Patologias Tropicais, Porto Velho, Rondônia